CLINICAL TRIAL: NCT00800579
Title: A Randomised, Double-blind, Placebo-controlled Trial to Assess the Safety, Tolerability and Pharmacokinetics of GS-9411 in Healthy Male Volunteers
Brief Title: Trial to Assess the Safety, Tolerability and Pharmacokinetics of GS-9411 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Thomas O'Riordan, MD, Gilead Sciences, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-221-0101
Record Dates: First submitted 2008-11-21; First posted 2008-12-02 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; CF; mucociliary clearance; amiloride; ENaC; ENaC Inhibitor; airway hydration; epithelial sodium channel inhibitor
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): GS-9411 0.6 mg
  Interventions: Drug: GS-9411
- 2 (Experimental): GS-9411 1.2 mg
  Interventions: Drug: GS-9411
- 3 (Experimental): GS-9411 2.4 mg
  Interventions: Drug: GS-9411
- 4 (Placebo Comparator): Inhaled volume-matched sterile saline placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-9411 — Inhaled GS-9411 dissolved in sterile saline
  Arms: 1; 2; 3
Drug: Placebo — Inhaled volume-matched placebo in sterile saline
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of escalating doses of GS-9411 in healthy male volunteers. GS-9411 is a sodium channel inhibitor, that may restore airway hydration and mucociliary clearance in the lung.

DETAILED DESCRIPTION:
GS-9411 is being evaluated as a potential therapy to improve airway hydration and mucociliary clearance in patients with cystic fibrosis. This study is evaluating the safety and tolerability of 3 dose levels of GS-9411 as an inhaled product, compared to a matched placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 to 45 years of age.
* No clinically important abnormal physical findings at screening.
* No clinically relevant abnormal lab results at screening.
* Normal (or abnormal but not clinically significant) ECG.
* Normal (or abnormal but not clinically significant) blood pressure (BP) and heart rate (HR).
* Body weight between 70 and 125 kg and body mass index (BMI) between 18 and 28 kg/m2, or outside range, but not clinically significant and agreed with sponsor and principal investigator.
* Able to communicate well with the investigator and to comply with the requirements of the entire study.
* Provision of written informed consent.
* Non-smokers of at least 6 months duration (< 10 pack year history) prior to study entry.
* Negative for drugs of abuse (including alcohol) at Screening and Day -5.
* Must be willing to abstain from alcohol and strenuous exercise during the 48-hour period prior to admission and while confined to the clinic.
* Forced expiratory volume in 1 second (FEV1) greater than or equal to 80% of predicted normal for age, gender, and height as per Hankinson et al1 at Screening and Pre-dose.
* Normal intraocular pressure between 10 and 22 mmHg.
* Male subjects who are sexually active must be willing to use effective barrier contraception (e.g., condom) during heterosexual intercourse from Baseline/Day 0 through completion of the study and continuing for at least 30 days from date of last dose of study drug.
* Male subjects must refrain from sperm donation from Day 1 through completion of the study and continuing for at least 30 days from the date of last dose of study drug.

Exclusion Criteria:

* Administration of any investigational drug in the period 0 to 12 weeks before entry to the study.
* A need for any medication during the period 0 to 5 days before entry to the study, except those deemed by the principal investigator/clinical investigator not to interfere with the outcome of the study.
* Existence of any surgical or medical condition which, in the judgment of the clinical investigator, might interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Presence or history of allergy requiring treatment. Hay fever is allowed unless it is active or has required treatment within the previous 2 months.
* Donation or loss of greater than 400 mL of blood in the period 0 to 12 weeks before entry to the study.
* Serious adverse reaction or hypersensitivity to any drug.
* Presence or history of any pulmonary diseases (e.g., asthma, emphysema, chronic bronchitis, cystic fibrosis, bronchiectasis).
* Consumption of drugs and/or herbal preparations capable of inducing hepatic enzyme metabolism (e.g., barbiturates, rifampicin, carbamazepine, phenytoin, primidone, or St. John's Wort) or enzyme-inhibiting agents (e.g., cimetidine) or similar drugs within 30 days (or 5 half-lives of inducing/inhibiting agent, whichever is longer) of enrollment in this study.
* Major surgery within 6 months of the start of this study.
* Subjects who have experienced a significant upper or lower respiratory tract infection within the 6 weeks prior to admission.
* Subjects with significant history of respiratory, renal, hepatic, cardiovascular (including history of systemic hypertension requiring therapy), metabolic, neurological, hematological, gastrointestinal, cerebrovascular, or other significant medical illness or disorder which, in the judgment of the investigator, may interfere with the study or require treatment which may affect the evaluation of efficacy and safety of the study drug.
* Subjects with elevated liver enzyme concentrations.
* Haemoglobin level < 130 g/L taken at Screening and at Pre-dose.
* Plasma potassium > 5 mEq/L taken at Screening and at Pre-dose.
* Poor venous access.
* Intraocular pressure > 21 mm Hg

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of 3 escalating doses of GS-9411 in healthy male volunteers | 11 Days

SECONDARY OUTCOMES:
To assess pharmacokinetics of GS-9411 and its metabolites | 11 Days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hodsman, MD, Principal Investigator — Nucleus Network Ltd
Locations (1):
- Nucleus Network Ltd., Melbourne, Victoria, Australia